CLINICAL TRIAL: NCT00942305
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study of the Safety, Tolerability and Ability of CMX001 to Prevent or Control CMV Infection in R+ Hematopoietic Stem Cell Transplant Recipients
Brief Title: Study of CMX001 to Prevent/Control Cytomegalovirus Infection in R+ Hematopoietic Stem Cell Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CMX001-201
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Cytomegalovirus Infection
Keywords: Allogeneic stem cell transplant; CMV seropositive (R+); transplant
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — brincidofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): * Cohort 1 = 40 mg of matching placebo administered once weekly (QW)
  * Cohort 2 = 100 mg of matching placebo administered QW
  * Cohort 3 = 200 mg of matching placebo administered QW
  * Cohort 4 = 200 mg of matching placebo administered twice weekly (BIW)
  * Cohort 4A = 100 mg of matching placebo administered BIW
  Interventions: Drug: Placebo
- Brincidofovir (Experimental): * Cohort 1 = 40 mg brincidofovir (BCV) administered once weekly (QW)
  * Cohort 2 = 100 mg BCV administered QW
  * Cohort 3 = 200 mg BCV administered QW
  * Cohort 4 = 200 mg BCV administered twice weekly (BIW)
  * Cohort 4A = 100 mg BCV administered BIW
  Interventions: Drug: Brincidofovir

INTERVENTIONS:
Drug: Brincidofovir — Subjects received their first dose of study drug of brincidofovir (BCV) within 30 (+5) days post-transplant and were treated through Week 13 post-transplant.
  Other Names: BCV; CMX001
  Arms: Brincidofovir
Drug: Placebo — Subjects received their first dose of study drug within 30 (+5) days post-transplant and were treated through Week 13 post-transplant.
  Matching placebo administered for each cohort.
  Arms: Placebo

SUMMARY:
This was a multicenter, randomized, double-blind, placebo-controlled, dose-escalation study of brincidofovir (BCV) administered orally once or twice weekly for up to 11 weeks. Dosing was initiated immediately following engraftment (between Days 14-30 post-transplant) to prevent/control cytomegalovirus (CMV) infection or prevent disease in R+ hematopoietic stem cell transplant (HCT) recipients.

DETAILED DESCRIPTION:
This was to be a 2-part study. Part 1 was a randomized, double-blind, placebo-controlled, dose-escalation study of multiple doses of oral brincidofovir (BCV) in R+ hematopoietic stem cell transplant (HCT) recipients. In Part 2, one of the dose levels administered in Part 1 was to be tested against placebo to evaluate the statistical significance of BCV as a therapy for preventing progression of cytomegalovirus (CMV) infection or preventing CMV disease. The first 3 dose-escalating cohorts in Part 1 were to include 32 subjects within each cohort (24 randomized to receive oral BCV and 8 randomized to receive placebo in a 3:1 ratio) for a total of 96 planned subjects. Following completion of the first 3 cohorts and subsequent safety review of the data, up to an additional 3 cohorts of 32 subjects each could have been enrolled. Two additional cohorts (labeled Cohort 4 and Cohort 4A) beyond the initial 3 cohorts were actually enrolled in Part 1 of the study. Following the safety and antiviral activity analyses of the 5 cohorts in Part 1 and the number of subjects enrolled in each of those cohorts, Part 2 of the study was not conducted.

ELIGIBILITY:
Inclusion Criteria

For inclusion into the study, all prospective subjects were required to fulfill all of the following criteria (as applicable):

1. Were aged ≥18 years. Males must have been able and willing to use adequate contraceptive methods throughout the treatment and follow-up phases of the study.
2. Were cytomegalovirus (CMV) seropositive before allogeneic hematopoietic stem cell transplantation (HCT) (i.e., R+ subjects).
3. Were less than 30 days post qualifying transplant.
4. Had evidence of engraftment before randomization and receiving their first dose of study drug.
5. Were able to ingest and absorb oral medication (in the judgment of the investigator and based on lack of significant gastrointestinal [GI] events).
6. Were willing and able to understand and provide written informed consent.
7. To the best of his or her knowledge, were willing and able to participate in all required study activities for the duration of the study.

Exclusion Criteria

Subjects meeting any of the following exclusion criteria were to be excluded from participation in the study:

1. Females who were pregnant or currently nursing.
2. Had a body mass index >35 kg/m2. [Note: This criterion was removed per Protocol Amendment 2 dated 27 August 2010.]
3. Had hypersensitivity to cidofovir (CDV) or brincidofovir.
4. Recipients for whom the current, predose clinical course of CMV infection suggested that the investigator would not be able to withhold treatment for CMV for a minimum of 5, but preferably 7 days following the subject's first dose of study drug.
5. Received any of the following:

   * Ganciclovir, valganciclovir, foscarnet or CDV within 14 days prior to enrollment;
   * Any anti-CMV therapy following transplantation (including Cytogam®1);
   * Any CMV vaccine;
   * Any investigational drug with antiviral activity against double-stranded DNA (dsDNA) viruses within 14 days prior to enrollment. [Note: An investigational drug was defined as a drug that was not approved for any indication by the Food and Drug Administration.]; or
   * Any other investigational drug (i.e., those without any "anti-dsDNA virus" activity; e.g., anti-influenza compounds) within 14 days prior to enrollment without the prior written consent of the medical monitor. The use of investigational drugs in certain circumstances was added per Protocol Amendment 1 dated 15 January 2010.
6. Received high dose acyclovir (>2000 mg total oral daily dose or >5 mg/kg intravenously 3 times daily) or valacyclovir (Valtrex; >3000 mg total daily dose) at the time of dosing.
7. Were diagnosed with active CMV disease within 6 months prior to enrollment; patients with CMV DNAemia requiring intervention with antiviral therapy at the time of enrollment.
8. Were HIV positive; patients with active hepatitis C virus (HCV) or hepatitis B virus (HBV) infection as evidenced by plasma levels of HCV RNA or HBV DNA, respectively.
9. Received another allogeneic HCT within the past 2 years, other than the qualifying HCT.
10. Had renal insufficiency as evidenced by glomerular filtration rate (GFR) <30 mL/min.
11. Had a current diagnosis of hypotony, uveitis, or retinitis or any intraocular pathology that would predispose the subject to any one of these conditions.
12. Had hepatic dysfunction as evidenced by alanine aminotransferase or aspartate aminotransferase >5 x the upper limit of normal (ULN) or direct bilirubin >2.5 x the ULN.
13. Had any of the following active autoimmune disorders: myasthenia gravis, Addison's disease, Wegener's granulomatosis, primary biliary cirrhosis, bullous pemphigoid, autoimmune hemolytic anemia, autoimmune hepatitis, multiple sclerosis, Goodpasture's syndrome, idiopathic thrombocytopenic purpura, lupus erythematosus, dermatomyositis, polymyositis, or vasculitis.
14. Had active solid tumor malignancies with the exception of basal cell carcinoma or the condition under treatment (e.g., lymphomas).
15. Had 1 or more episode of hyperglycemic coma or diabetic ketoacidosis within the 6 months prior to enrollment.
16. Had cardiovascular disease which, in the opinion of the investigator, would interfere with the conduct of the study.
17. Had Grade 3 or 4 graft versus host disease of the GI tract; subjects with any GI disease that would, in the judgment of the investigator, preclude the subject from taking or absorbing oral medication (e.g. clinically active Crohn's disease, ischemic colitis, moderate or severe ulcerative colitis, or any condition expected to require abdominal surgery during the course of study participation).
18. Any other condition including abnormal laboratory values that would have, in the judgment of the investigator, put the subject at increased risk for participating in the trial, or interferes with the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Moores UCSD Cancer Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Brigham and Womens Hospital, Division of Infectious Disease, Boston, Massachusetts
  - University of Michigan Medical School, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mt. Sinai School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center Oncology, The Bronx, New York
  - UNC Health Care Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists - Intermountain Healthcare, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lanier ER, Foster S, Brundage T, Chou S, Prichard MN, Kleiboeker S, Wilson C, Colville D, Mommeja-Marin H. Analysis of Mutations in the Gene Encoding Cytomegalovirus DNA Polymerase in a Phase 2 Clinical Trial of Brincidofovir Prophylaxis. J Infect Dis. 2016 Jul 1;214(1):32-5. doi: 10.1093/infdis/jiw073. Epub 2016 Mar 3. PMID 26941282
- [Result] Marty FM, Winston DJ, Rowley SD, Vance E, Papanicolaou GA, Mullane KM, Brundage TM, Robertson AT, Godkin S, Mommeja-Marin H, Boeckh M; CMX001-201 Clinical Study Group. CMX001 to prevent cytomegalovirus disease in hematopoietic-cell transplantation. N Engl J Med. 2013 Sep 26;369(13):1227-36. doi: 10.1056/NEJMoa1303688. PMID 24066743
- [Derived] Tippin TK, Morrison ME, Brundage TM, Mommeja-Marin H. Brincidofovir Is Not a Substrate for the Human Organic Anion Transporter 1: A Mechanistic Explanation for the Lack of Nephrotoxicity Observed in Clinical Studies. Ther Drug Monit. 2016 Dec;38(6):777-786. doi: 10.1097/FTD.0000000000000353. PMID 27851688
- See also: Analysis of Mutations in Gene Encoding Cytomegalovirus DNA Polymerase in a Phase 2 Clinical Trial of Brincidofovir Prophylaxis — http://pubmed.ncbi.nlm.nih.gov/26941282/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note: While a total of 239 subjects were enrolled, 1 center was excluded from analysis due to concerns about investigator/site compliance with the study protocol. This center had enrolled 9 subjects: 5 subjects who received brincidofovir (BCV) in Cohort 1, 2 subjects who received placebo in Cohort 1, and 2 subjects who received BCV in Cohort 2.
Groups:
- Cohort 1 BCV: 40 mg brincidofovir (BCV) administered once weekly
- Cohort 1 Placebo; Cohort 2 Placebo; Cohort 3 Placebo: Placebo administered once weekly (QW)
- Cohort 2 BCV: 100 mg brincidofovir (BCV) administered once weekly
- Cohort 3 BCV: 200 mg brincidofovir (BCV) administered once weekly
- Cohort 4 BCV: 200 mg brincidofovir (BCV) administered twice weekly (BIW)
  Note: This dose was reduced to 200 mg BCV once weekly for ongoing subjects in this cohort following the recommendation of the Data and Safety Monitoring Board. No new subjects were enrolled into this cohort following the decision to reduce the dose.
- Cohort 4 Placebo; Cohort 4a Placebo: Placebo administered twice weekly (BIW)
- Cohort 4a: 100 mg brincidofovir (BCV) administered twice weekly (BIW)
Period: Overall Study
Arm/Group | Cohort 1 BCV | Cohort 1 Placebo | Cohort 2 BCV | Cohort 2 Placebo | Cohort 3 BCV | Cohort 3 Placebo | Cohort 4 BCV | Cohort 4 Placebo | Cohort 4a | Cohort 4a Placebo
Started | 30 | 10 | 29 | 10 | 39 | 14 | 30 | 10 | 50 | 17
Completed | 7 | 5 | 14 | 4 | 14 | 9 | 6 | 5 | 25 | 7
Not Completed | 23 | 5 | 15 | 6 | 25 | 5 | 24 | 5 | 25 | 10

BASELINE CHARACTERISTICS:
Population: Note: While a total of 239 subjects were enrolled, 1 center was excluded from analysis due to concerns about investigator/site compliance with the study protocol. This center had enrolled 9 subjects: 5 subjects who received brincidofovir (BCV) in Cohort 1, 2 subjects who received placebo in Cohort 1, and 2 subjects who received BCV in Cohort 2.
Groups:
- Cohort 1 BCV: 40 mg brincidofovir (BCV) administered once weekly (QW)
- Cohort 2 BCV: 100 mg brincidofovir (BCV) administered once weekly (QW)
- Cohort 3 BCV: 200 mg brincidofovir (BCV) administered once weekly (QW)
- Cohort 4a BCV: 100 mg brincidofovir (BCV) administered twice weekly (BIW)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 BCV | Cohort 1 Placebo | Cohort 2 BCV | Cohort 2 Placebo | Cohort 3 BCV | Cohort 3 Placebo | Cohort 4 BCV | Cohort 4 Placebo | Cohort 4a BCV | Cohort 4a Placebo | Total
Number analyzed (Participants) | 25 | 8 | 27 | 10 | 39 | 14 | 30 | 10 | 50 | 17 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.02) | 56.8 (10.12) | 51.7 (10.13) | 53.5 (11.08) | 49.5 (12.75) | 47.9 (14.05) | 50.4 (11.47) | 52.2 (14.76) | 48.8 (12.74) | 46.1 (12.14) | 50.7 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 1 | 10 | 5 | 17 | 9 | 12 | 3 | 24 | 7 | 98
  Male | 15 | 7 | 17 | 5 | 22 | 5 | 18 | 7 | 26 | 10 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant CMV Infection
Description: The primary efficacy endpoint was a binomial outcome of failure to prevent cytomegalovirus (CMV) infection defined as CMV DNAemia >200 copies/mL obtained at the time of the last treatment with study drug or diagnosis of CMV disease at some point during the treatment phase.
Time Frame: Randomization to Week 8 post-treatment (~19 weeks)
Population: Modified Intent-to-Treat Population, which included all randomized subjects who took at least 1 dose of study treatment and who had at least 1 efficacy evaluation following baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 BCV | Cohort 1 Placebo | Cohort 2 BCV | Cohort 2 Placebo | Cohort 3 BCV | Cohort 3 Placebo | Cohort 4 BCV | Cohort 4 Placebo | Cohort 4a BCV | Cohort 4a Placebo
Number analyzed (Participants) | 25 | 8 | 27 | 10 | 39 | 14 | 30 | 10 | 50 | 17
Participants | 13 | 4 | 6 | 4 | 12 | 4 | 7 | 3 | 5 | 7

ADVERSE EVENTS:
Arm/Group | Cohort 1 BCV | Cohort 1 Placebo | Cohort 2 BCV | Cohort 2 Placebo | Cohort 3 BCV | Cohort 3 Placebo | Cohort 4 BCV | Cohort 4 Placebo | Cohort 4a BCV | Cohort 4a Placebo
Serious Adverse Events (participants affected / at risk) | 12/25 | 4/8 | 10/27 | 6/10 | 19/39 | 6/14 | 21/30 | 3/10 | 30/50 | 8/17
Other Adverse Events (participants affected / at risk) | 25/25 | 8/8 | 27/27 | 9/10 | 39/39 | 14/14 | 30/30 | 10/10 | 50/50 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 BCV (N=25) | Cohort 1 Placebo (N=8) | Cohort 2 BCV (N=27) | Cohort 2 Placebo (N=10) | Cohort 3 BCV (N=39) | Cohort 3 Placebo (N=14) | Cohort 4 BCV (N=30) | Cohort 4 Placebo (N=10) | Cohort 4a BCV (N=50) | Cohort 4a Placebo (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 10 | 0 | 5 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2 | 3 | 0 | 1 | 2 | 2 | 2
Cholecytitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 12 | 0 | 15 | 2
Acute graft versus host disease in intestine (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Acute graft versus host disease in liver (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Acute graft versus host disease in skin (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BK virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Citrobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Serratia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Viral haemorrhagic cystitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Bacteria stool identified (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Espstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 BCV (N=25) | Cohort 1 Placebo (N=8) | Cohort 2 BCV (N=27) | Cohort 2 Placebo (N=10) | Cohort 3 BCV (N=39) | Cohort 3 Placebo (N=14) | Cohort 4 BCV (N=30) | Cohort 4 Placebo (N=10) | Cohort 4a BCV (N=50) | Cohort 4a Placebo (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 2 | 2 | 2 | 1 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 4 | 1 | 4 | 0 | 4 | 2 | 10 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 1 | 0 | 1 | 5 | 0 | 7 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 2 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid margin crusting (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myodesopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 2 | 0 | 5 | 1 | 11 | 0 | 13 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1 | 1 | 3 | 0 | 2 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 8 | 4 | 13 | 4 | 21 | 2 | 26 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 4 | 2 | 1 | 0 | 4 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 4 | 0 | 2 | 0 | 2 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 5 | 1 | 11 | 4 | 11 | 3 | 17 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 6 | 2 | 6 | 4 | 8 | 1 | 22 | 3
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 3 | 0 | 1 | 1 | 3 | 1 | 2 | 1 | 1 | 2
Chills (General disorders) | 1 | 1 | 0 | 1 | 3 | 3 | 0 | 1 | 2 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 3 | 0 | 5 | 3 | 0 | 1 | 9 | 3
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 0 | 5 | 1 | 3 | 2 | 3 | 2 | 8 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 3 | 7 | 1 | 2 | 2 | 10 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 5 | 0 | 3 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 24 | 2 | 32 | 6
Acute graft versus host disease in intestine (Immune system disorders) | 2 | 0 | 5 | 1 | 6 | 2 | 0 | 0 | 0 | 0
Acute graft versus host disease in skin (Immune system disorders) | 4 | 2 | 3 | 3 | 7 | 0 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 0
Aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
BK virus infection (Infections and infestations) | 1 | 0 | 4 | 1 | 3 | 1 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 3 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 2 | 2 | 4 | 2 | 2 | 3 | 2 | 1
Cytomegalovirus viraemia (Infections and infestations) | 10 | 2 | 4 | 2 | 7 | 3 | 5 | 0 | 6 | 4
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 6 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 5 | 0
Proctitis herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0
Viral haemorrhagic cystitis (Infections and infestations) | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 0 | 2 | 0 | 10 | 0 | 9 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 1 | 7 | 0 | 5 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 5 | 0 | 3 | 2 | 2 | 0 | 7 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 4 | 0
Blood urea increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Echocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 4 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 1
Immunosuppressant drug level increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 0
Weight decreased (Investigations) | 3 | 0 | 4 | 0 | 0 | 3 | 1 | 2 | 6 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 5 | 1 | 3 | 1 | 5 | 2 | 9 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 4 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 8 | 0 | 9 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 3 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 2 | 1 | 5 | 1 | 5 | 2 | 8 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 3 | 1 | 2 | 2 | 1 | 0 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0 | 7 | 1 | 2 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 4 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 3 | 0 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 4 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 3 | 3 | 1 | 0 | 3 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 0 | 3 | 2 | 3 | 0 | 4 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 3 | 0 | 4 | 1
Headache (Nervous system disorders) | 0 | 1 | 3 | 0 | 3 | 2 | 4 | 1 | 3 | 3
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Peropheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 3 | 0 | 3 | 0 | 2 | 0 | 2 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 3 | 2 | 3 | 1 | 2 | 0 | 3 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 1 | 1 | 2 | 0 | 3 | 0 | 3 | 2 | 4 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 2 | 0 | 5 | 1 | 2 | 0 | 9 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 2 | 3 | 2 | 3 | 1 | 1 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 2 | 1 | 2 | 0 | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 3 | 1 | 0 | 0 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 4 | 1 | 0 | 2 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 4 | 2 | 4 | 1 | 1 | 0 | 5 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 1 | 4 | 2 | 6 | 1 | 6 | 3
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 3 | 2 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Cholitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Acute graft versus host disease in liver (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Serratia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Viral tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 18 months after the end of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment. Institution publication may be delayed up to an additional 45 days to allow Sponsor to seek patent protection.